CLINICAL TRIAL: NCT07022795
Title: Effectiveness of an Ecological Momentary Assessment Intervention to Reduce Masticatory Muscle Activity in Individuals at Risk for Temporomandibular Disorders
Brief Title: Behavioral Interventions for Controlling Oral Behaviors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Iacopo Cioffi, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 46622
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Temporomandibular Disorders (TMD); Bruxism; Masseter
Keywords: awake bruxism; temporomandibular disorders; masseter; oral behaviors; surface electromyography; tooth clenching
MeSH Terms: conditions — Temporomandibular Joint Disorders; Bruxism

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The operator performing the data analysis will be blinded to the research dataset through dataset masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Group A
  Interventions: Behavioral: Educational video only
- Standard of care combined with an ecological momentary assessment intervention (Experimental): Group B
  Interventions: Behavioral: Educational video combined with daily surveys

INTERVENTIONS:
Behavioral: Educational video combined with daily surveys — Participants will receive the same educational intervention as those in the other arm and will also undergo an ecological momentary assessment (EMA) intervention. This will involve receiving multiple messages per day on their mobile phones, each linking to an online survey designed to capture real-time data on their current oral behaviors. The intervention aims to increase participants' awareness of these behaviors by prompting them to reflect on and report them throughout the day.
  Arms: Standard of care combined with an ecological momentary assessment intervention
Behavioral: Educational video only — Participants will be provided with an educational video on recognizing and managing oral behaviors such as clenching, prolonged tooth contact, and keeping the jaw tense, etc.
  The goal is to increase awareness and promote behavior change to reduce strain to the masticatory muscles and the temporomandibular joint.
  Arms: Standard of care

SUMMARY:
Ecological momentary assessment (EMA) interventions via mobile devices can be implemented to monitor an individual's negative health behaviors in real-time, increase awareness, and assist patients in overting those behaviors. In recent years, EMA interventions have been used to improve patients' awareness of specific oral behaviors, such as tooth clenching or awake bruxism, which can produce excessive forces on the muscles of mastication and lead to or exacerbate symptoms of temporomandibular disorders (TMD). Yet, whether EMA interventions are effective in reducing oral behaviors and masticatory muscle activity in the short- and long-term, or whether they are more effective than patient education remains unclear.

In this randomized clinical trial, we aim to test the effects of a 1-week EMA intervention combined with structured information on masticatory muscle activity and determine whether a combined approach including an EMA intervention and structured information is more effective in reducing masticatory muscle activity than structured information alone.

Our study will have a significant impact on orofacial pain clinical research as it will provide clinically relevant measures which could inform multimodal approaches for the management of painful TMD.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) are the most common cause of nondental orofacial pain (1) and the second most frequent painful musculoskeletal (MSK) disorder after chronic low back pain (2). TMD affect 1/6 Canadians, mostly women (3). Painful TMD can affect the muscles of mastication and/or the temporomandibular joints (TMJs, i.e., the jaw joints), and are characterized primarily by spontaneous pain, or pain associated with jaw function, and TMJ sounds (e.g., clicking) (4). TMD pain affecting the muscles of mastication (TMD myalgia; mTMD) is the most common TMD (5). MTD mostly affect the two major muscles of mastication, i.e. the masseter and the temporalis. As in other painful MSK conditions, TMD cause considerable personal suffering, and pose a significant economic burden (6). In the USA ~$4 billion are spent annually, with >17.8 million lost work days/year for every 100 million working adults (7). Notably, ~85% of the cost of treating TMD is associated with clinical management of chronic mTMD. Despite the high prevalence of TMD, more than 30% of patients report pain for at least 5 years after treatment, regardless the treatment they had received (8) which suggests that treatments for TMD are ineffective. Consensus has been achieved in that conservative management strategies should be preferred over more invasive treatment approaches, such as prolonged pharmacological treatments or opioid use, which result in significant adverse effects that impact significantly on the quality of life of patients (9). Of importance, both laboratory and epidemiological studies indicated that oral behaviors - for example, awake bruxism, a stress-coping behavior characterized by repetitive or sustained tooth clenching(10)- might harm the muscles of mastication or the jaw joint (the temporomandibular joint, TMJ) by way of producing excessive forces to which these structures are exposed, potentially leading to, or exacerbating symptoms of TMD (11). Therefore, patient education focused on reducing the frequency of oral behaviors or awake bruxism has proven to be an effective first-line approach towards mTMD management (12-13). Notably, highly frequent oral behaviors and awake bruxism also can increase the risk of prosthetic failure (e.g., damage to restorations or crowns/bridges (14), which poses a financial burden to patients. As such, behavioral interventions aiming at monitoring and reducing oral behaviors could benefit a significant proportion of patients submitted to prosthetic rehabilitations as well.

Ecological momentary assessment (EMA) involves real-time and repeated assessments of phenomena (e.g., frequency of behaviors, mood states, symptoms etc.) over a period of time in naturalistic or ambulatory environments (15). In medicine and dentistry, EMA has been used to assist in the diagnosis of chronic pain disorders, including facial pains, such as migraine (6-18). By collecting specific features of a patient's symptoms (e.g., pain duration, intensity, location) on portable devices in real time, it is possible to develop temporal trajectories of those features, which can assist in achieving a clinical diagnosis, or study relationships between clinical symptoms and other variables (e.g., those related with lifestyle or the local environment).

EMA has been previously used in clinical research studies to assess the prevalence of oral behaviors in healthy individuals or in those affected with TMD, and to study facial pain temporal trajectories in individuals with chronic pain (16-17) (19-21). EMA studies have confirmed that individuals with TMD have more frequent oral behaviors than healthy controls (21-23). In the clinical realm, it is widely accepted that EMA interventions could be implemented to reduce the frequency of oral behaviors in patients with TMD pain. In fact, by providing real-time data and reports on an individual's frequency of oral behaviors, EMA could assist patients in monitoring and overcoming those oral behaviors (24). Notably, patient education through structured information about the detrimental effects of oral behaviors on the muscles of mastication and the temporomandibular joint (TMJ) has also been shown to be effective in reducing masticatory muscle activity and temporomandibular disorder (TMD) pain in the short term (12). Yet, whether EMA is more effective than structured information in reducing oral behaviors and masticatory muscle activity remains unclear. Although EMA interventions are conservative in nature, they can significantly disrupt an individual's daily life, as the EMA methodology requires the use of portable devices (such as tablets or mobile phones) to prompt an individual multiple times a day at random. As such, there is a need to understand whether this intervention is effective. Importantly, we lack information on the long-term effectiveness of EMA interventions. Of concern, individuals in specific job categories may be prevented from undergoing EMA interventions.

In this randomized clinical trial, we aim 1) to test the effects of a 1-week EMA intervention combined with structured information on the activity of the masseter muscle in individuals reporting highly frequent self-reported oral behaviors (high risk of TMD) (25), and 2) to determine whether a combined approach including an EMA intervention and structured information is more effective in reducing the activity of the masseter than structured information alone. We hypothesize that 1) EMA intervention + structured information will reduce the frequency of non-functional muscle contraction episodes (assessed with portable electromyography) only in the short-term, i.e., 1 week after its completion, and after one month, and 2) that EMA intervention combined with structured information will not be more effective than structured information alone.

REFERENCES. 1. Benoliel R. & Sharav Y. Curr Pain Headache Rep 2010; 14:33-40; 2. National Institute of Dental And Craniofacial Research NIDCR, 2020; 3. Locker D. & Slade G. Community Dent Oral Epidemiol. 1988;16:310-313; 4. Schiffman E. et al. J Oral Facial Pain Headache. 2014; 28:6-27; 5. Manfredini D. et al. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011; 112:453-462; 6. Slade G. et al. J Dent Res. 2016; 95: 1084-1092; 7. Maixner W. et al. J Pain. 2011;12: T4-8.e11-12. 13; 8. Fricton J.R. et al. Advances in Pain Research and Therapy; Orofacial Pain and Temporomandibular Disorders. New York: Raven Press; 1995; 9. National Academies of Sciences Engineering and Medicine. Temporomandibular Disorders: Priorities for Research and Care. Washington: The National Academies Press, 2020; 10. Manfredini D. & Lobbezoo F. J Orofac Pain. 2009;23:153-166; 11. Cioffi I. et al. Clin Oral Investig. 2017; 21:1139-1148; 12. Donnarumma V. et al. J Oral Facial Pain Headache. 2022:36-48; 13. Durham J. J Oral Rehabil. 2016;43: 929-936; 14. Johansson A. J Prosthodont Res. 2011;55: 127-36; 15. Shiffman S. 2008;4:1-32; 16. Edefonti V. Community Dent Oral Epidemiol. 2012;40 Suppl 1:56-64; 17. Cioffi I, J Oral Rehabil. 2017;44:333-339; 18. Thomas JG. Cephalalgia. 2016;36:1228-1237. 19. Kaplan SE & Ohrbach R. J Oral Facial Pain Headache. 2016;30:107-19; 20. Michelotti A. et al. J Dent Res. 2005;84:644-8; 21. Câmara-Souza M.B. et al. J Clin Med. 2023; 7;12:501; 22. Glaros A.G. et al. J Am Dent Assoc. 2005;136:451-8; 23. Glaros A.G. et al. Cranio. 2005;23:188-93; 24. Glaros A.G. et al. Appl Psychophysiol Biofeedback. 2007;32:149-54; 25. Ohrbach R. et al. J Pain. 2013;14(12 Suppl):T33-50; 26. Markiewicz M.R., et al. J Orofac Pain. 2006;20:306-16; 27. Ohrbach R. Eur J Oral Sci. 2008;116:438-44; 28. Cioffi I. et al. Clin Oral Investig. 2017;21:1139-1148. 29. Imbriglio T.V. et al. Headache. 2020;60:2389-2405; 30. Prasad S. et al. Clin Oral Investig. 2021;25:5049-5059; 31. Lou T et al.. Am J Orthod Dentofacial Orthop. 2021;159(1):e25-e33; 32. Chow J.C. & Cioffi I. Clin Oral Investig. 2019; 23:1653-1661

ELIGIBILITY:
Individuals reporting a score greater than or equal to 25 on the oral behavior checklist (OBC). The OBC is a self-report questionnaire used to assess the frequency of various daytime and sleep-related oral behaviors, such as teeth clenching, grinding, and jaw tension.

It helps identify habits that may contribute to temporomandibular disorders (TMD) and orofacial pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of oral behaviors | after one week intervention
  Frequency of electromyographic (EMG) activity periods greater than 5 and 10% of participants' maximum voluntary contraction, measured using ambulatory EMG.

SECONDARY OUTCOMES:
Duration of oral behaviors | after one week intervention
  Duration of electromyographic (EMG) activity periods greater than 5 and 10% of participants' maximum voluntary contraction, measured using ambulatory EMG

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared with third parties, in accordance with the currently approved research ethics protocol.